CLINICAL TRIAL: NCT01700777
Title: Effet de la réadaptation Sur Les déficiences, Limitations d'activité et Restriction de la Participation Des Enfants présentant Des lésions Neurologiques Non-évolutives (Infirmes Moteurs cérébraux).
Brief Title: Bimanual Training in Children With Hemiplegia With Lower Limb and Postural Stimulation (HABIT & Leg)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Scientific collaborator, Institute of Neuroscience UCL, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHMG-IONS-862010
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Congenital Hemiplegia
Keywords: bimanual training; lower limb; intensive rehabilitation; regular rehabilitation; hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Neurological Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive rehab group (Experimental): A group of children will beneficiate of "HABIT-ILE" treatment in an intensive way (camp) for 90h.
  Interventions: Other: "HABIT-ILE"
- Regular treatment group (Active Comparator): A group of children with hemiplegic cerebral palsy will beneficiate from conventional training at a regular frequency (1 to 6 hours / week) for 90hours.
  Interventions: Other: "HABIT-ILE"

INTERVENTIONS:
Other: "HABIT-ILE" — 90 h of training with "HABIT-ILE", in an intensive rehabilitation camp compared with a regular therapy program (groups are crossed-over afterwards).
  Other Names: Bimanual training, HABIT, neurorehabilitation

SUMMARY:
A randomized control trial of "HABIT-ILE" therapy compared with regular / conventional intervention (same amount of hours). The protocols have been developed on the basis of bimanual therapy (HABIT) developed at Columbia University.

DETAILED DESCRIPTION:
A randomized control trial of "HABIT-ILE" therapy at intensive frequency contrasted with regular frequency intervention. The protocols have been developed on the basis of bimanual therapy (HABIT) developed at Columbia University. The intervention takes place either in a 2 weeks day and night camp, either in regular/conventional intervention (1 to 5 hours a week). Children of all groups will benefit from 90h of intensive treatment (children in regular frequency will be crossed over afterwards to benefit from HABIT-ILE. Both in the camp and the regular interventions, there is at least one therapist for each child.

ELIGIBILITY:
Inclusion Criteria:

* willingness to enter the research program and the testing procedures

Exclusion Criteria:

* uncontrolled epilepsy
* upper limb injections in the upper limb during the last six months / or intend to receive during the training period

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Impairment, disability, participation | 4 years
  The 3 WHO main domains will be investigated. Impairments will be investigated through force, sensory and manipulation testing (including manipulation with mechanical device). Analysis of lower limb is also included in the protocol. Disabilities will be tested through video-taped assessments and questionnaires. Participation will be assessed through questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, PhD, Principal Investigator — Institute of Neurosciences, UCL; Corinne Bleyenheuft, MD, Principal Investigator — Cliniques Universitaires de Mont-Godinne
Locations (1):
- Institute of Neurosciences, UCL, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Derived] Araneda R, Dricot L, Ebner-Karestinos D, Paradis J, Gordon AM, Friel KM, Bleyenheuft Y. Brain activation changes following motor training in children with unilateral cerebral palsy: An fMRI study. Ann Phys Rehabil Med. 2021 May;64(3):101502. doi: 10.1016/j.rehab.2021.101502. Epub 2021 Mar 22. PMID 33647530
- [Derived] Bleyenheuft Y, Dricot L, Ebner-Karestinos D, Paradis J, Saussez G, Renders A, De Volder A, Araneda R, Gordon AM, Friel KM. Motor Skill Training May Restore Impaired Corticospinal Tract Fibers in Children With Cerebral Palsy. Neurorehabil Neural Repair. 2020 Jun;34(6):533-546. doi: 10.1177/1545968320918841. Epub 2020 May 14. PMID 32407247
- [Derived] Bleyenheuft Y, Arnould C, Brandao MB, Bleyenheuft C, Gordon AM. Hand and Arm Bimanual Intensive Therapy Including Lower Extremity (HABIT-ILE) in Children With Unilateral Spastic Cerebral Palsy: A Randomized Trial. Neurorehabil Neural Repair. 2015 Aug;29(7):645-57. doi: 10.1177/1545968314562109. Epub 2014 Dec 19. PMID 25527487